CLINICAL TRIAL: NCT01884194
Title: Morphological Analysis of the Pineal Gland in Pediatric Retinoblastoma Patients Using Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Thi Thai Hien Pham, doctoral candidate, Charite University, Berlin, Germany
Other Study IDs: RTB_0305_outcome
Record Dates: First submitted 2013-05-24; First posted 2013-06-21 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Retinoblastoma; Pineoblastoma
Keywords: retinoblastoma; pineoblastoma
MeSH Terms: conditions — Retinoblastoma; Pinealoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retinoblastoma patients: patients with diagnosed retinoblastoma
- non-retinoblastoma patients: aged matched control cohort without the diagnosis of ocular or brain tumor

SUMMARY:
MRI is useful for diagnosing pinealoblastoma in retinoblastoma patients

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of retinoblastoma
* brain MRI available

Exclusion Criteria:

* insufficient quality of brain MRI

Ages: 1 Day to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients with retinoblastoma
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Malignancy criteria of pineal gland | clinical follow-up 1-year after baseline imaging
  size of pineal gland solid or cystic component (all at baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Charite Hospital Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Pham TT, Siebert E, Asbach P, Willerding G, Erb-Eigner K. Magnetic resonance imaging based morphologic evaluation of the pineal gland for suspected pineoblastoma in retinoblastoma patients and age-matched controls. J Neurol Sci. 2015 Dec 15;359(1-2):185-92. doi: 10.1016/j.jns.2015.10.046. Epub 2015 Oct 28. PMID 26671110